CLINICAL TRIAL: NCT03623269
Title: Posterior Approach to Total Shoulder Arthroplasty: A Data Analysis on Patients Undergoing the Posterior Approach to Total Shoulder Arthroplasty
Brief Title: Posterior Approach to Total Shoulder Arthroplasty
Acronym: pTSA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Orthopaedic Research & Innovation Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ORIF.005
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Total Shoulder Arthroplasty; Osteo Arthritis Shoulders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: posterior approach to total shoulder arthroplasty — The posterior approach to total shoulder arthroplasty approaches the patient from the back of the shoulder and spares the rotator cuff.

SUMMARY:
The purpose of this study is to evaluate preoperative objective measurements and operative objective measurements to determine if there is any effect to postoperative outcomes. Patients who were 18 years old or greater at the time of surgery were followed clinically and radiographically to determine best practice and optimal treatment and technique, risk and rate of complication, and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. >18 years of age
3. Underwent posterior approach to total shoulder arthroplasty by Dr. Michael Greiwe at St. Elizabeth Healthcare

Exclusion Criteria:

1. Non-English speaking
2. <18 years of age
3. Loose bone in the anterior recess of the shoulder
4. Severe arthritis with significant bony deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible patients of the principal investigator receiving the posterior approach to total shoulder arthroplasty for any indication at our institution between September 1, 2016 and October 31, 2017 were evaluated and included in the data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
recovery | preoperative to 6 months postoperatively
  American shoulder and elbow score (ASES) with a range from 0-100, with 0 being worst outcome and 100 being best outcome
recovery | preoperative to 6 months postoperatively
  Simple Shoulder Test score (SST) with a range from 0-12 with 12 being the best score and 0 being the worst score.
recovery | preoperative to 6 months postoperatively
  range of motion
complications | 6 months postoperative
  percent of complications

CONTACTS AND LOCATIONS:
Overall Officials: R M Greiwe, MD, Principal Investigator — The Orthopaedic Research & Innovation Foundation
Locations (1):
- The Orthopaedic Research & Innovation Foundation, Edgewood, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided